CLINICAL TRIAL: NCT00901771
Title: A Non-randomized, Case Series Study of the Effectiveness of Provent Treatment of Obstructive Sleep Apnea Patients Who Are Non-compliant or Minimally Adherent With Positive Airway Pressure Therapy
Brief Title: Study of Provent Treatment of Obstructive Sleep Apnea in Patients Who Are Non-compliant With CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Hospital, Chesterfield, Missouri (Other)
Collaborators: Ventus Medical, Inc. (Industry)
Responsible Party: James K. Walsh, Ph.D., Sleep Medicine and Research Center at St. Luke's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ventus C020
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep; Sleep Apnea, Obstructive; OSA; OSAH
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Provent — This is a non-randomized, single-arm, case series study. All subjects will receive Provent device.

SUMMARY:
The primary objective of the proposed investigation is to evaluate the efficacy of the Provent device in a sample of OSA patients who have either refused or been non-adherent with PAP treatment. Both initial efficacy (evaluated after approximately one week with Provent) and efficacy after approximately 5 weeks in patients who demonstrate initial efficacy will be assessed. A secondary objective is to assess adherence with Provent treatment during the 5-week evaluation period.

ELIGIBILITY:
Inclusion Criteria:

* Current signs and symptoms consistent with a diagnosis of OSA in the opinion of the study physician
* Rejection of PAP treatment or minimally adherent with PAP treatment
* Use of the Provent device for a specified amount of time each night during three consecutive nights of the trial period
* AHI > 15, or AHI > 10 with evidence of CMS-recognized symptoms or co- morbidities, on screening/baseline PSG
* Investigator believes that subject can benefit from OSA treatment
* Subject understands and is willing and able to comply with study requirements

Exclusion Criteria:

* Use of any device that interferes with nasal or oral breathing
* Persistent blockage of one or both nostrils which prevents airflow in one or both nostrils
* Any chronic sores or lesions on the inside or outside of the nose
* Chronic use of nasal decongestants other than nasal steroids
* History of allergic reaction to acrylic-based adhesives (such as those found in BAND-AIDS®)
* Current acute upper respiratory (including nasal, sinus, or middle ear) inflammation or infection or perforation of the tympanic membrane (may be re-considered for participation after the acute episode resolves)
* History of frequent and/or poorly treated severe nasal allergies or sinusitis which may interfere with the ability to use Provent
* Severe respiratory disorders (including respiratory muscle weakness, bullous lung disease, bypassed upper airway, pneumothorax, pneumomediastinum, etc.).
* Pathologically low blood pressure.
* Narcolepsy, idiopathic hypersomnolence, chronic insomnia, restless legs syndrome, REM sleep behavior disorder or any other diagnosed or suspected sleep disorder other than OSA that could affect the likelihood of apneas/hypopneas during a PSG.
* Periodic limb movement arousal index (PLMAI) > 10 on the screening/baseline PSG.
* Current use of diurnal or nocturnal supplemental oxygen
* Currently working night or rotating shifts
* Consumption of > 10 caffeinated beverages per day (approximately 1000 mg per day)
* History of severe cardiovascular disease, including New York Heart Association Class III or IV heart failure, coronary artery disease with angina or myocardial infarction in the past 6 months, stroke in the past 6 months
* History of cardiac rhythm disturbance (defined as a 5-beat run of sustained ventricular tachycardia or bradycardia if < 30 beats per min for a 10-second run or previously undiagnosed and untreated atrial fibrillation or Mobitz II or third-degree heart block)
* Current psychiatric disorder with psychotic features.
* Pregnant or trying to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Week 1 AHI as compared to Screening/Baseline AHI | 1 week

SECONDARY OUTCOMES:
Week 5 AHI as compared to Screening/Baseline AHI | 5 weeks
Minutes with SaO2 <90%: Week 5 vs. Screening/Baseline | 5 weeks
Epworth Sleepiness Scale: Week 5 vs. Baseline | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James K Walsh, Ph.D., Principal Investigator — Sleep Medicine and Research Center at St. Luke's Hospital
Locations (1):
- Sleep Medicine and Research Center at St. Luke's Hospital, Chesterfield, Missouri, United States